CLINICAL TRIAL: NCT06093295
Title: Using Non-invasive Brain Stimulation to Modulate Injury Risk Biomechanics Among Individuals With and Without a Concussion History
Brief Title: Non-invasive Brain Stimulation and Injury Risk Biomechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PROJECT00007759
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Concussion, Mild
Keywords: concussion; repetitive transcranial magnetic stimulation; mild traumatic brain injury; biomechanics; reaction time; theta burst stimulation
MeSH Terms: conditions — Brain Concussion | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The researchers will employ a single-blinded cross-over study design.
Who Masked: Participant
Masking Description: The researchers will employ a single-blinded cross-over study design. The participant will not know which day the participant receives the true (experimental) or control (placebo) repetitive transcranial magnetic stimulation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Left Dorsolateral Prefrontal Cortex (experimental) (Experimental): This is the experimental condition where participants will receive theta burst stimulation to the left dorsolateral prefrontal cortex.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (Theta Burst Stimulation)
- Vertex (control) (Placebo Comparator): This is the control condition where participants will receive theta burst stimulation to the vertex.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (Theta Burst Stimulation)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (Theta Burst Stimulation) — The repetitive transcranial magnetic stimulation device will generate successive magnetic pulses to the left dorsolateral prefrontal cortex (experimental condition) and the vertex (control condition).
  The theta burst stimulation protocol is as follows:
  * Total stimulation time ~190 seconds
  * Intensity: 80% of active motor threshold
  * 2 seconds train, repeated every 10 seconds
  * In every 2-second train, 3 pulses of stimulation are delivered at 50 Hz, repeated every 200 milliseconds (i.e., 5 Hz) for a total of 600 pulses

SUMMARY:
The goal of this clinical trial is to test the effects of repetitive transcranial magnetic stimulation (theta burst stimulation) on movement biomechanics (jump landing) among individuals with and without a concussion history. The main question it aims to answer is if theta burst stimulation to the left dorsolateral prefrontal cortex improves single- and dual-task jump landing reaction time and jump landing biomechanics compared to a control site (vertex) for individuals with and without a concussion history.

Participants will be asked to perform a jump landing before and after the experimental (left dorsolateral prefrontal cortex) and control (vertex) theta burst stimulation protocol. The researchers will compare individuals with and without a concussion history to see if the effects differ between groups.

DETAILED DESCRIPTION:
The overall goal of the project is to determine how repetitive transcranial magnetic stimulation (theta burst stimulation) influences movement among individuals with and without a concussion history. The purpose of this study is prevention via improving injury risk biomechanics to reduce the risk of future musculoskeletal injury.

Participants will complete 2 testing sessions separated by a minimum of 7 days.

During the first testing session, participants will complete single-task serial subtraction, single- and dual-task jump landing, and a theta burst stimulation intervention. The jump landing will be completed before and after theta burst stimulation and under single- and dual-task (serial 7s) conditions. During the second testing session, participants will complete the jump landing before and after theta burst stimulation under single- and dual-task (serial 7s) conditions.

On both testing sessions, the symptom checklist and Tampa Scale of Kinesiophobia 11 (TSK-11) will be administered upon arrival to the lab (after informed consent on day 1), and immediately after repetitive transcranial magnetic stimulation. The Godin Leisure Activity Questionaire will be administered on both days before the jump landing. The NASA Task Load index will be administered on both days immediately after the completion of every cognitive and motor task.

At the end of the second day of testing, the participants will be asked which day the participants believed the participants received the experimental and control conditions of the theta burst stimulation intervention.

This is a single-blinded cross-over design study. The participants will be unaware of when the participants receive the true (experimental) and control (placebo) theta burst stimulation intervention. Experimental (left dorsolateral prefrontal cortex) and control (vertex) conditions will be counterbalanced for the concussion history group. The control group will be matched to their respective concussion history group counterpart's counterbalanced order.

ELIGIBILITY:
Inclusion Criteria:

All participants

* self-report to be physically active at least 90 minutes per week
* aged 18-35 years old
* self-report cleared for sports and physical activity

Concussion history group

- self-report experiencing a concussion with the National Institute of Health common data element form

No concussion history group - self-report not experiencing a concussion with the National Institute of Health common data element form

Exclusion Criteria:

All Participants

* self-report attention deficit disorder and/or attention deficit hyperactivity disorder
* self-report uncorrected vision problems (not included color blindness)
* self-reported history of neurological disease
* self-reported history of seizures/syncope or family history of epilepsy
* self-reported history of frequent severe headaches or migraine.
* self-reported history of respiratory or heart disease.
* self-reported structural brain lesions (e.g., stroke)
* self-reported increased intracranial pressure, such as after infarctions or trauma.
* self-reported currently using antidepressants, neuroleptic medication, medication that lowers seizure threshold, or any other medication that would interfere with testing.
* self-reported currently experiencing a high fever (day of testing; >102.9 degrees)
* self-reported currently undergoing immunosuppressive therapy
* pregnancy
* metal anywhere in the head (except the mouth).
* any electronic implant, such as a cardiac pacemakers, cochlear implant, or deep brain stimulator.
* any implanted medication pump or intracardiac lines.
* self-report not being cleared for sport/physical activity by a medical practitioner (i.e., must be cleared by a medical practitioner to participate if the participant had previous traumatic musculoskeletal injury)
* students working directly in the PI's lab (concussion laboratory, biomechanics laboratory)
* NCAA athletes

Concussion history group

- ≥13 symptom severity on the Sport Concussion Assessment Tool (22 total symptoms are graded on a scale of 0-6. Any symptom with a score >0 [1-6], is summed to get symptom severity).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Reaction Time | Immediately before and immediately after both theta burst stimulation conditions.
  The time between the audible buzzer and the when sacral marker moves >3 cm in the sagittal or transverse plane.
Knee Flexion Angle | Immediately before and immediately after both theta burst stimulation conditions.
  The angle of the shank relative to the thigh in the sagittal plane (deg).
Knee Abduction Angle | Immediately before and immediately after both theta burst stimulation conditions.
  The angle of the shank relative to the thigh in the frontal plane (deg).
Hip Flexion Angle | Immediately before and immediately after both theta burst stimulation conditions.
  The angle of the thigh relative to the pelvis in the sagittal plane (deg).
Hip Adduction Angle | Immediately before and immediately after both theta burst stimulation conditions.
  The angle of the thigh relative to the pelvis in the frontal plane (deg).
Trunk Flexion Angle | Immediately before and immediately after both repetitive theta burst stimulation conditions.
  The angle of the trunk relative to the lab in the sagittal plane (global axis system; deg).
Trunk Lateral Bending Angle | Immediately before and immediately after both theta burst stimulation conditions.
  The angle of the trunk relative to the lab in the frontal plane (global axis system; deg)

SECONDARY OUTCOMES:
NASA Task Load Index | After every cognitive condition during the jump landing on both the experimental and control theta burst stimulation days.
  The NASA Task Load Index is abbreviated NASA-TLX. The NASA-TLX is a self-reported assessment to assess the workload and effort of a given task. There are 6 domains (mental demand, physical demand, temporal demand, performance, effort, and frustration) each scored on a scale of 0 to 20. A score of 0 indicates "very low", and a score of 20 indicates "very high". The raw scores will be summed together for analysis. Higher scores indicate greater workload and effort. The NASA-TLX will be analyzed as a continuous variable ranging from 0-120.
Tampa Scale of Kinesiophobia 11 | Immediately before and immediately after the experimental and control theta burst stimulation.
  The Tampa Scale of Kinesiophobia 11 (TSK-11) is a self-reported assessment to assess the participant's fear of movement. The TSK-11 ranges on a scale from 11-44. Higher scores on the TSK-11 indicate a greater fear of movement. TSK-11 will be analyzed as a continuous variable ranging from 11-44.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Lynall, Phd, ATC, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Master data files will be available upon reasonable request.

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Ngetich R, Jin D, Li W, Song B, Zhang J, Jin Z, Li L. Enhancing Visuospatial Working Memory Performance Using Intermittent Theta-Burst Stimulation Over the Right Dorsolateral Prefrontal Cortex. Front Hum Neurosci. 2022 Mar 17;16:752519. doi: 10.3389/fnhum.2022.752519. eCollection 2022. PMID 35370586
- [Background] Shumski EJ, Anderson MN, Oh J, Schmidt JD, Lynall RC. Computerized and functional reaction time in varsity-level female collegiate athletes with and without a concussion history. J Sci Med Sport. 2023 Mar;26(3):189-194. doi: 10.1016/j.jsams.2023.02.008. Epub 2023 Mar 3. PMID 36906428
- [Background] Lynall RC, Blackburn JT, Guskiewicz KM, Marshall SW, Plummer P, Mihalik JP. Reaction Time and Joint Kinematics During Functional Movement in Recently Concussed Individuals. Arch Phys Med Rehabil. 2018 May;99(5):880-886. doi: 10.1016/j.apmr.2017.12.011. Epub 2018 Jan 11. PMID 29337022
- [Background] Said S, Gozdzik M, Roche TR, Braun J, Rossler J, Kaserer A, Spahn DR, Nothiger CB, Tscholl DW. Validation of the Raw National Aeronautics and Space Administration Task Load Index (NASA-TLX) Questionnaire to Assess Perceived Workload in Patient Monitoring Tasks: Pooled Analysis Study Using Mixed Models. J Med Internet Res. 2020 Sep 7;22(9):e19472. doi: 10.2196/19472. PMID 32780712
- [Background] Chimenti RL, Post AA, Silbernagel KG, Hadlandsmyth K, Sluka KA, Moseley GL, Rio E. Kinesiophobia Severity Categories and Clinically Meaningful Symptom Change in Persons With Achilles Tendinopathy in a Cross-Sectional Study: Implications for Assessment and Willingness to Exercise. Front Pain Res (Lausanne). 2021 Sep 1;2:739051. doi: 10.3389/fpain.2021.739051. eCollection 2021. PMID 35295417
- [Background] Woby SR, Roach NK, Urmston M, Watson PJ. Psychometric properties of the TSK-11: a shortened version of the Tampa Scale for Kinesiophobia. Pain. 2005 Sep;117(1-2):137-44. doi: 10.1016/j.pain.2005.05.029. PMID 16055269